CLINICAL TRIAL: NCT02952105
Title: Identification of Ventricular Fibrillation and Optimization of Defibrillation During Chest Compression of CPR: A Multiple Study of Cardiac Arrest Patients in China.
Brief Title: Identification of Ventricular Fibrillation and Optimization of Defibrillation During CPR
Acronym: IVFOD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: Peking Union Medical College Hospital (Other); Jinhua Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UST20161009
Record Dates: First submitted 2016-10-30; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Arrest; Identify of Electrocadiac Rhythm
Keywords: cardiac arrest; identify of electrocardiac rhythm; ventricuar fibrillation; defibrillation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- defibrillation patients: shockable rhythm, defibrillated
- non defibrillation patients: non-shockable rhythm, non defibrillated

SUMMARY:
It's so important to recognize ventricular fibrillation in cardiac arrest and defibrillation early. At the same time Research findings have identified high-quality CPR with minimum interruption is critical to the success of defibrillation therapy. Both the guidelines by American Heart Association and the guidelines by European Resuscitation Council emphasize the importance of minimizing interruptions in chest compressions, specifically, duration of the pre-shock and post-shock pauses. So AHA indicate that there will be a new algorithm of VF during chest compression, which has high sensitivity and specificity. And the investigators can identify VF and defibrillate earlier.

The aim of this study is to verify that if Sherlock algorithm of Philips MRx monitor/defibrillator can identify shockable rhythms during chest compression accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac arrest patients
2. The length from cardia arrest to be rescued is less than 10 minutes
3. age≥14
4. Complied with ethical requirements
5. signing the informed consent form.

Exclusion Criteria:

1. DNR
2. Pregnant women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cardiac arrest patients aged more than 14 years
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Sherlock algorithm of Philips MRx monitor/defibrillator in identify ventricular fibrillation. | 04/10/2016-10/01/2017
How long it is advanced that the first time Sherlock algorithm identified VF than the true time VF was recognized. | 04/10/2016-10/01/2017
Comparasion of no-flue time between true scene and assumed scene that useing Sherlock algorithm. | 04/10/2016-10/01/2017

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhong Yu, Doctor, Study Chair — Peking Union Medical College Hospital; Guoxiu Zhang, Bachelor, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Mingwei Huang, Bachelor, Study Director — Jinhua Central Hospital
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided